CLINICAL TRIAL: NCT01576913
Title: Music Pacing in Pediatric Exercise Testing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Principal Investigator, Gal Raz-Dubnov MD, MSc, senior physician, Sheba Medical Center
Allocation: Randomized | Model: Crossover | Masking: Single
Other Study IDs: SHEBA-12-9340-GDR-CTIL
Record Dates: First submitted 2012-04-11; First posted 2012-04-13 (Estimated); Last update posted 2014-11-25 (Estimated); Status verified 2014-11

CONDITIONS: Exercise Testing With Music Pacing
Keywords: exercise testing; music; VO2 max

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Music pacing (Active Comparator): Exercise testing with music pacing
  Interventions: Other: Music listening
- No music pacing (No Intervention): Exercise testing without music pacing

INTERVENTIONS:
Other: Music listening — Listening to tempo music while cycling in an exercise test
  Arms: Music pacing

SUMMARY:
Study hypothesis: Music pacing improves the quality of exercise testing in children.

Children tend to cycle in a non-constant pace during exercise testing, which might make the test less reliable.

20 boys will perform two exercise tests on a cycle ergometer. One test will be done with constant tempoed music, and the other without. Different parameters will be checked including pedaling cadence, aerobic fitness, level of work load obtained.

ELIGIBILITY:
Inclusion Criteria:

* male sex
* currently and generally healthy

Exclusion Criteria:

* presence of chronic disease/ medication use
* BMI above 85%
* trained/competitive cyclists

Ages: 8 Years to 12 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2012-04; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
peak VO2 | end of the exercise test, approx.10 minutes
  peak Vo2 is the maximal oxygen consumption obtained during the exercise test, reflecting the level of aerobic fintess

SECONDARY OUTCOMES:
peak power | exercise test duration, approx.10 minutes
  maximal power obtained at the end of the exercise test
anaerobic threshold | exercise test duration, approx.10 minutes
  point of increase in anaerobic metabolism
rating of perceived exertion | exercise test duration, approx.10 minutes
  scale of perceived effort
mechanical efficiency | exercise test duration, approx.10 minutes
  oxygen consumption per work load
cadence | exercise test duration, approx.10 minutes
  pedaling rate

CONTACTS AND LOCATIONS:
Overall Officials: Gal Dubnov-Raz, MD, MSc, Principal Investigator — Sheba Medical Center
Locations (1):
- Sheba_Medical_Center, Ramat Gan, Israel